CLINICAL TRIAL: NCT00634452
Title: A Phase 1, Open-label, Dose-escalation, Multidose Study of MDX-1401 Administered Weekly for 4 Weeks in Patients With CD30-positive Refractory/Relapsed Hodgkin's Lymphoma
Brief Title: Phase 1 Study of MDX-1401 in Patients With CD30-positive Refractory/Relapsed Hodgkin's Lymphoma
Acronym: MDX1401-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX1401-01; CA213-001 (Other: BMS)
Record Dates: First submitted 2008-02-26; First posted 2008-03-13 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hodgkin's Lymphomas
Keywords: Hodgkin's; Cancer; bi-measurable disease; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Neoplasms; Lymphoma | interventions — MDX-1401

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDX-1401 (Experimental): MDX-1401 iv at various doses
  Interventions: Biological: MDX-1401

INTERVENTIONS:
Biological: MDX-1401 — IV weekly for 4 weeks

SUMMARY:
To establish the safety and tolerability profile of MDX-1401 in patients with relapsed or refractory Hodgkin's Lymphoma (HL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD30-positive HL by immunohistochemistry or flow cytometry
* Must have failed or relapsed following second line chemotherapy or radiation or failed/relapsed following autologous stem cell transplant
* Bi-measurable disease
* ECOG Performance Status of 0 - 2
* Meet all screening laboratory values

Exclusion Criteria:

* Previous treatment with any other anti-CD30 antibody
* History of allogeneic transplant
* Any tumor lesion greater than or equal to 10 cm in diameter
* Any active or chronic significant infection
* Underlying medical condition which will make the administration of MDX- 1401 hazardous
* Concomitant corticosteroids, chemotherapy, investigational agents, other anti-HL biologics, or radiation therapy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Profile | Two years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Day 50
Tumor response assessment | Two year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (6):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - ClinWorks Cancer Research Center, Charlotte, North Carolina
  - Scott and White Memorial Hospital and Clinic, Temple, Texas
  - West Virginia University, Morgantown, West Virginia